CLINICAL TRIAL: NCT07116226
Title: Learning How to Implement and Use a Ketogenic Diet to Improve Mental Health
Acronym: LIVE IT~LAUNCH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Deanna Kelly, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HP-00113852
Record Dates: First submitted 2025-06-09; First posted 2025-08-11 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Medical Keto Diet
Keywords: Medical Ketogenic Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical Keto Mastery Class (Experimental)
  Interventions: Other: Medical Keto Education Program

INTERVENTIONS:
Other: Medical Keto Education Program — 4 hour asynchronous educational class

SUMMARY:
The goal of the study is to implement a team-based "train the trainer" group approach by providing participants education and the opportunity for self-implementing a medical ketogenic diet study for 4 weeks.

The overarching goal of the program is for those participating to be able to initiate the diet in clinical and research settings with greater competence.

The study has two parts:

1. Mastery Class (Education, Q & A)
2. 4 Week Open Label LIVE IT ketogenic diet participation with private and group consultation (optional)

DETAILED DESCRIPTION:
There will be two parts to assist with a train the trainer approach: 1) an educational component (4-hour mastery class, 2 Q&A 1.5 hours) with related materials and 2) an open label cohort study providing the opportunity for participants to attempt the medical ketogenic diet within a group for 4 weeks with private and group counseling.

By participating in a 4-week self-implemented diet within a group setting our hope is to increase competence in implementing the diet and monitoring its success with KetoMojo. Secondarily, those who participate in the cohort study may have improvements in their own physical health and mental well-being.

After the 4 hour mastery class is completed an additional two weeks is given prior to the group keto diet starting to ensure all dietician meetings are completed.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-74 years
* Not currently on a ketogenic diet
* No prior experience in successfully implementing a medical ketogenic diet for self
* Clinician, researcher or clinical or research team member

Exclusion Criteria:

* Age 18-74 years
* Body mass index > 18.5
* Not currently on a ketogenic diet (Self report)
* No prior experience in successfully implementing a medical ketogenic diet for self (Self report)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in individual competence in understanding the nutritional aspects and food selection of a medical keto diet. Competence will be measured by pre- and post-education and post- LlVE IT experience (optional) | 12 weeks
  This will be assessed with16 items answerable along a Visual Analog scale each with scores from 0-100mm with higher scores demonstrating better competence.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, PharmD, BCPP, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Maryland Psychiatric Research Center (MPRC), Catonsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No